CLINICAL TRIAL: NCT02569671
Title: Immediate Placement of the Straumann® Bone Level Tapered Implant With Early Loading in Single Tooth Gaps in the Maxilla and Mandible Compared to Delayed Placement
Brief Title: Bone Level Tapered Multi-Center Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 01/14
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Tooth Loss
Keywords: Dental Implants, Single-Tooth
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Immediate Placement - Test (Other): Straumann Bone Level Tapered Implant - Immediate Placement - Implant is placed at the time of tooth extraction to replace a single tooth.
  Interventions: Device: Straumann Bone Level Tapered Implant - Immediate Placement
- Delayed Placement - Control (Other): Straumann Bone Level Tapered Implant - Delayed Placement - Implant is placed after 16-18 weeks of healing to replace a single tooth.
  Interventions: Device: Straumann Bone Level Tapered Implant - Delayed Placement

INTERVENTIONS:
Device: Straumann Bone Level Tapered Implant - Immediate Placement — Immediate placement of a Straumann Bone Level Tapered Dental Implant for replacement of a singe tooth.
  Arms: Immediate Placement - Test
Device: Straumann Bone Level Tapered Implant - Delayed Placement — Delayed placement of a Straumann Bone Level Tapered Dental Implant for replacement of a singe tooth.
  Arms: Delayed Placement - Control

SUMMARY:
The aim of this randomized, controlled, multi-center study is to assess the clinical and radiographic outcomes of using a Straumann® Bone Level Tapered implant for immediate implantation following extraction of a tooth in the pre-molar and anterior region of the maxilla and mandible (test) compared to the outcomes of placing this implant in healed sites (control).

DETAILED DESCRIPTION:
The primary objective is to demonstrate that the change in mean peri-implant marginal bone level changes (mesial and distal) from loading to 12 months post-loading of the test treatment will not be worse than the control treatments.

The secondary objectives of the study are to assess differences in clinical and radiographic outcomes between the test and control treatments at 12 months post-loading by looking at implant success and survival, buccal bone dimensional changes, implant stability, soft tissue changes, subject satisfaction, and adverse events.

An additional objective is to assess long-term differences in clinical and radiographic outcomes, as measured in the primary and secondary objectives, over the span of two, three, four, and five years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form before any study related procedures
* Subjects must be males or females who are a minimum of 18 years of age
* Subjects who are in need of a single tooth extraction in the pre-molar or anterior region of the maxilla or mandible (ADA tooth positions 4-13 and 20-29) and replacement with a dental implant.
* Implants must be placed either immediately in an extraction socket or placed in a healed site (greater than 4 months healing) which has not been previously grafted.
* Planned site for implant must have a natural tooth both mesially and distally in the adjacent tooth positions
* Subjects must have opposing dentition (natural teeth, fixed or removable restorations)
* There must be sufficient bone at the implant site to achieve primary stability
* Subjects must be committed to the study and the required follow-up visits
* Subjects must be in good general health as assessed by the Investigator

Exclusion Criteria:

* Subjects with a systemic disease that would preclude dental implant surgery
* Subjects with any contraindications for oral surgical procedures
* Subjects with mucosal diseases (e.g., erosive lichen planus) in the localized area around the study implant site
* Subjects with a history of local irradiation therapy in the head/neck area
* Subjects with any untreated endodontic lesions or untreated periodontal disease adjacent to the implant site
* Subjects receiving, or having a history of receiving, intravenous or subcutaneous antiresorptive agents, such as bisphosphonates
* Subjects with severe bruxing, parafunctional habits, or temporomandibular joint dysfunction
* Any implant sites where there will be a buccal dehiscence greater than 3 mm or there will be a fenestration of the implant
* Subjects with inadequate oral hygiene or who are unmotivated for adequate home care
* Subjects who have physical or mental handicaps that would interfere with the ability to perform adequate oral hygiene
* Subjects who are pregnant or intending to become pregnant during the duration of the study
* Subjects who are heavy smokers (defined as >10 cigarettes per day or >1 cigar per day) or chew tobacco
* Subjects who abuse alcohol or drugs
* Subjects who have undergone administration of any investigational device within 30 days of enrollment in the study
* Subjects with conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2025-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David L. Cochran, DDS, PhD, MS, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (3):
- United States (3):
  - UCLA School of Dentistry, Los Angeles, California
  - Center for Implant Dentistry, University of Florida, Gainesville, Florida
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Placement - Test | Delayed Placement - Control
Started (65 subjects were screened before randomization) | 26 | 27
Completed | 23 | 23
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: Male or female subjects aged 18 years or older required a single tooth extraction in the premolar or anterior region of the maxilla or mandible and met the inclusion criteria but not the exclusion or withdrawal criteria were included in the study population. During the surgical procedure, participants were allowed to have multiple teeth extracted and/or multiple implants inserted, but only one implant was designated as the study implant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Placement - Test | Delayed Placement - Control | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 54.5 (13.7) | 57.0 (15.0) | 55.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 9 | 13 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 17 | 20 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Mean Crestal Bone Level Change
Description: mean crestal bone level at 12 months - mean crestal bone level at implant loading (baseline) = Change in crestal bone level
Time Frame: Measured at implant loading (10-12 weeks after implant surgery) and 12 months post-loading
Population: 65 subjects were screened, 11 were screen failures and 1 pre-randomizatio lost to follow-up.
  From the 53 subjects randomized (ITT group), 50 subjects (25 in the test, 25 in the control group) received the study treatment (mITT).
  Among mITT group, 5 lacked primary analysis measurements: 3 control, 2 test.
  Test group (N=23) had 1 lost follow-up, 1 lost implant post-op. Control group (N=22) had 1 baseline measurement missing, 2 lost implants post-restoration.
Measure: Mean (Standard Deviation); unit: Change in Mean crestal bone levels (mm)
Groups:
- Immediate Placement (Test Group): Straumann Bone Level Tapered Implant - Immediate Placement - Implant is placed at the time of tooth extraction to replace a single tooth.
- Delayed Placement (Control Group): Straumann Bone Level Tapered Implant - Delayed Placement - Implant is placed after 16-18 weeks of healing to replace a single tooth.
Arm/Group | Immediate Placement (Test Group) | Delayed Placement (Control Group)
Number analyzed (Participants) | 23 | 22
Change in Mean crestal bone levels (mm) | 0.5 (0.6) | 0.5 (0.7)
Statistical Analysis 1: Comparison: Immediate Placement (Test Group) vs Delayed Placement (Control Group); The null hypothesis for the primary analysis is that the difference between the mean change in crestal bone levels for the treatment and control groups is at least the non-inferiority margin (indicating inferior bone gain). Rejection of the null hypothesis indicates the observed data supports the alternative hypothesis that the difference between the mean change in crestal bone levels for the treatment and control groups; Test type: Non-Inferiority — is less than the non-inferiority margin (indicating non-inferior bone gain). The hypotheses associated with the primary analysis are defined as: H0: µc - µs ≥ δ H1: µc - µs < δ where µc is the mean change in crestal bone levels from implant loading to 12 months post-implant loading for the treatment group, µs is the mean change for the control group, and δ is the 0.5 mm non-inferiority margin. The hypotheses will be tested using a one-sided t-test with a 5% significance level; p = .950, t-test, 1 sided — SD for both test and control group is 0.5 mm, A difference between groups of ≥ 0.5 mm is considered clinically significant, The difference between the treatment groups is expected to be 0 mm, Statistical test will be one-sided 5% significance level; The hypotheses will be tested using a one-sided t-test with a 5% significance level; Mean Difference (Final Values) = 0.5, Standard Deviation 0.5 — The hypotheses will be tested using a one-sided t-test with a 5% significance level; The change in mean bone level from implant loading to 12-month follow-up was calculated. Change in crestal bone levels was calculated as the crestal bone level at 12-months post implant loading minus crestal bone level at implant loading

2. Secondary Outcome: Implant Success and Survival
Description: Control group N-25 Test group N=24
  Survival and success was assessed by the dimensions below as noted by Buser.
  * Absence of persistent subjective complaints, such as pain, foreign body sensation, and/ or dysesthesia
  * Absence of a recurrent peri-implant infection with suppuration
  * Absence of mobility
  * Absence of a continuous radiolucency around the implant
Time Frame: 12 months post-loading
Population: 65 subjects were screened, 11 were screen failures and 1 pre-randomizatio lost to follow-up.
  From the 53 subjects randomized (ITT group), 50 subjects received the study treatment (mITT).
  Test group (N=24) had 1 lost follow-up Control group (N=25)
Measure: Count of Participants; unit: Participants
Groups:
- Immediate Placement (=Test Group): Straumann Bone Level Tapered Implant - Immediate Placement - Implant is placed at the time of tooth extraction to replace a single tooth.
- Delayed Placement (=Control Group): Straumann Bone Level Tapered Implant - Delayed Placement - Implant is placed after 16-18 weeks of healing to replace a single tooth.
Arm/Group | Immediate Placement (=Test Group) | Delayed Placement (=Control Group)
Number analyzed (Participants) | 24 | 25
Participants
  Lost Implant | 1 | 2
  surviving and successful implant at 12 months | 23 | 23

3. Secondary Outcome: Buccal Bone Dimensional Changes
Description: Buccal bone dimensional changes were measured on images recorded on cone beam computed tomography (CBCT). The average of the following measurement locations is reported as outcome variable:
  1) mesial to distal; 2) distal-buccal; 3) mid-buccal; 4) mesial-buccal; 5) distal-lingual; 6) mid-lingual; 7) mesial-lingual.
Time Frame: Measured at Implant loading and at screening and 12 months post-loading
Population: At Implant Loading - Test group N=23, Control N=23 At 12 month Follow Up - Test group N=22, Control N=23
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Immediate Placement (=Test Group) | Delayed Placement (=Control Group)
Number analyzed (Participants) | 22 | 22
mm
  Mean Buccal Bone Dimensional Change at Implant loading | 2.1 (0.6) | 2.0 (0.5)
  Mean Buccal Bone Dimensional Change at 12 months post loading | 2.1 (0.7) | 1.8 (0.6)
Statistical Analysis 1: Comparison: Immediate Placement (=Test Group) vs Delayed Placement (=Control Group); All secondary effectiveness endpoints were planned to be summarized descriptively, and no hypothesis tests was planned; Test type: Non-Inferiority — Smaller bone dimensional thickness of the buccal plate measurements indicates less bone loss and better healing; p = 0.022, t-test, 1 sided; The hypotheses will be tested using a one-sided t-test with a 5% significance level; Mean Difference (Final Values) = 0.1, Standard Deviation 0.3

4. Secondary Outcome: Implant Measure as Measured by ISQ at Implant Surgery
Description: Implant stability as measured by ISQ held facial-lingual and held mesial-lingual.
  An Osstell device that uses the Resonance Frequency Analysis (RFA) method to determine implant stability and osseointegration was used in the study. The results were presented as an Implant Stability Quotient (ISQ) value of 1 - 100. The higher the ISQ, the more stable the implant. Additional information about the Osstell device can be found at www.osstell.com. Instructions on taking the measurements for this protocol will be provided in the Operation Manual. Two measurements were taken from two different angles at implant placement, implant loading, and final restoration.
Time Frame: Implant surgery: Immediate Placement for Test Group = implant is placed at the time of tooth extraction. Delayed Placement is Control Group= implant is placed after 16-18 weeks of healing
Population: Implant stability was measured by resonance frequency analysis implant surgery. 25 subject from each group (control and test) received an implant and had ISQ assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Placement (=Test Group) | Delayed Placement (=Control Group)
Number analyzed (Participants) | 25 | 25
Participants
  ISQ Value 1: Probe held facial-lingual: ISQ < 60 | 9 | 0
  ISQ Value 1: Probe held facial-lingual: ISQ 60 to 69 | 2 | 2
  ISQ Value 1: Probe held facial-lingual: ISQ ≥ 70 | 14 | 23
  ISQ Value 2: Probe held mesial-lingual: ISQ < 60 | 7 | 0
  ISQ Value 2: Probe held mesial-lingual: ISQ 60 to 69 | 4 | 1
  ISQ Value 2: Probe held mesial-lingual: ISQ ≥ 70 | 14 | 24

5. Secondary Outcome: Implant Stability as Measured by ISQ at Implant Loading
Description: Implant stability was measured by ISQ and probe held facial-lingual and held mesial-lingual.
  An Osstell device is an instrument that uses the Resonance Frequency Analysis (RFA) method to determine implant stability and osseointegration. The result is presented as an Implant Stability Quotient (ISQ) value of 1 - 100. The higher the ISQ, the more stable the implant. Additional information about the Osstell device can be found at www.osstell.com. Instructions on taking the measurements for this protocol will be provided in the Operation Manual. Two measurements will be taken from two different angles at implant placement, implant loading, and final restoration.
Time Frame: Implant Loading=implant surgery + 10 weeks (+/-3 weeks)
Population: 23 subjects from Test group and 24 from Control group had ISQ assessed at Implant Loading.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Placement (=Test Group) | Delayed Placement (=Control Group)
Number analyzed (Participants) | 23 | 24
Participants
  ISQ Value 1 Probe held facial-lingual measured at Implant Loading: ISQ < 60 | 0 | 1
  ISQ Value 1 Probe held facial-lingual measured at Implant Loading: ISQ 60 to 69 | 4 | 3
  ISQ Value 1 Probe held facial-lingual measured at Implant Loading: ISQ ≥ 70 | 19 | 20
  ISQ Value 2: Probe held mesial-lingual measured at Implant Loading: ISQ < 60 | 0 | 1
  ISQ Value 2: Probe held mesial-lingual measured at Implant Loading: ISQ 60 to 69 | 4 | 3
  ISQ Value 2: Probe held mesial-lingual measured at Implant Loading: ISQ ≥ 70 | 19 | 20

6. Secondary Outcome: Implant Stability as Measured by ISQ at Final Restoration
Description: as for outcome 5
Time Frame: Final Restoration: 10 weeks post-loading (± 2 weeks)
Population: 23 subjects from Test and 24 from Control group had ISQ assessed at Final Restoration visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Placement (=Test Group) | Delayed Placement (=Control Group)
Number analyzed (Participants) | 23 | 24
Participants
  ISQ Value 1: Probe held facial-lingual: ISQ < 60 | 1 | 1
  ISQ Value 1: Probe held facial-lingual: ISQ 60 to 69 | 3 | 1
  ISQ Value 1: Probe held facial-lingual: ISQ ≥ 70 | 19 | 22
  ISQ Value 2: Probe held mesial-lingual: ISQ < 60 | 0 | 1
  ISQ Value 2: Probe held mesial-lingual: ISQ 60 to 69 | 2 | 1
  ISQ Value 2: Probe held mesial-lingual: ISQ ≥ 70 | 21 | 22

7. Secondary Outcome: Change in Soft Tissue Measurements
Description: The following table illustrates a comparison between Soft Tissue Mean Changes Around the Implant for delayed and immediate placements, measured at final restoration (10 weeks post loading) and the 12-month mark post implant loading. The parameters assessed included: CLTm (length of crown from highest point of soft tissue to incisal edge of the adjacent mesial tooth), CLTd (length of crown from highest point of soft tissue to incisal edge of the adjacent distal tooth), CLI (length of the implant crown from highest point of the soft tissue margin to the incisal edge), IPm (distance from the top of the papilla to the incisal edge mesial of the implant crown), IPd (distance from the top of the papilla to the incisal edge distal of the implant crown)
Time Frame: Soft tissue measurements were taken and compared between the test and the control group at final restoration (10 weeks post loading) and 12 months (± 1 month) post implant loading (implant loading=implant surgery + 10 weeks (+/-3 weeks)).
Population: Measurements of soft tissue changes around the implant were recorded at both the time of final restoration (10 weeks post-loading) and the 12-month Follow-up (12 months post-loading). Specifically, 23 subjects from the Test group and 23 from the Control group had their soft tissue measurements changes assessed at 12 months follow-up (post-loading).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Immediate Placement (=Test Group) | Delayed Placement (=Control Group)
Number analyzed (Participants) | 23 | 23
mm
  Change in CLTm from final restoration to 12-month follow-up (mm) | -0.3 (1.9) | 0.1 (0.8)
  Change in CLTd from final restoration to 12-month follow-up (mm) | -0.2 (2.2) | 0.1 (1.1)
  Change in CLI from final restoration to 12-month follow-up (mm) | -0.4 (1.8) | -0.1 (0.8)
  Change in IPm from final restoration to 12-month follow-up (mm) | -0.5 (1.2) | -0.5 (1.5)
  Change in IPd from final restoration to 12-month follow-up (mm) | -0.7 (1.6) | -0.7 (1.6)

8. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction related to pain, crown's esthetic, and crown's function was assessed at 12 months post-loading using Visual Analog Scales (VAS). Satisfaction range between 0 to 100 with Excruciating and Not satisfied at all at zero point and Nonexistent and Extremely satisfied at the 100 point. The table summarizes pain, satisfaction with function and satisfaction with esthetics at 12-months post loading.
Time Frame: 12 months post-loading
Population: In each group, Test and Control, 25 subjects underwent implant placement, and Subject satisfaction related to pain, crown's esthetic, and crown's function was assessed using Visual Analog Scales (VAS).
  Specifically, 23 subjects from the Test group and 23 from the Subject satisfaction related to pain, crown's esthetic, and crown's function was assessed at 12 months post-loading using Visual Analog Scales (VAS).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Placement (=Test Group) | Delayed Placement (=Control Group)
Number analyzed (Participants) | 23 | 23
score on a scale
  Pain associated with implant crown | 5.9 (20.6) | 14.7 (33.8)
  Satisfaction with function | 97.9 (5.2) | 97.8 (6.6)
  Satisfaction with esthetics | 96.5 (6.1) | 96.3 (9.2)

9. Secondary Outcome: Number of Participants With Adverse Events and Adverse Device Effects Over 12 Months
Description: The frequency of adverse events and adverse device effects will be determined at 12 months post-loading and compared between the test and control arms. There were 38 total Adverse Events in 18 subjects out of 53 subjects. There were no SAEs related to procedure or device.
Time Frame: Measured at each study visit and throughout 12 months
Population: Over a 12-month period, 38 adverse events (AEs) were reported among 18 of the 53 study subjects. The randomization process assigned 26 subjects to the test group (=immediate placement) and 27 subjects to the control group (=delayed placement). No serious adverse events (SAEs) related to the procedure or device were observed.
Measure: Count of Participants; unit: Participants
Groups:
- Immediate Placement (=Test Group): Straumann Bone Level Tapered Implant - Immediate Placement (=Test Group) - Implant is placed at the time of tooth extraction to replace a single tooth.
- Delayed Placement (=Control Group): Straumann Bone Level Tapered Implant - Delayed Placement (=Control Group)- Implant is placed after 16-18 weeks of healing to replace a single tooth.
Arm/Group | Immediate Placement (=Test Group) | Delayed Placement (=Control Group)
Number analyzed (Participants) | 26 | 27
Participants
  Any Adverse Events | 6 | 12
  Adverse Device Effects | 2 | 4
  Device Related | 1 | 2
  Procedure Related | 2 | 3
  Serious Adverse Events | 2 | 4
  Serious Adverse Device Events | 0 | 0
  SAE Device Related | 0 | 0
  SAE Procedure Related | 0 | 0

ADVERSE EVENTS:
Time Frame: For the avoidance of doubt, all AE/SAEs as defined below, regardless of whether they are related to the investigational device, were collected , fully investigated and documented in the source document and appropriate case report form for all subjects from the time of the signing of the informed consent until the 60 months (post-loading) follow-up visit. An AE is defined as any untoward medical occurrence, unintended disease or injury, or any untoward clinical signs in subjects.
Description: An AE is defined as any untoward medical occurrence, unintended disease or injury, or any untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.
Groups:
- Immediate Placement (= Test Group): 26 Immediate Placement (= Test Group)
- Delayed Placement (= Control Group): 27 Delayed Placement (= Control Group)
Arm/Group | Immediate Placement (= Test Group) | Delayed Placement (= Control Group)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/26 | 4/27
Other Adverse Events (participants affected / at risk) | 8/26 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Placement (= Test Group) (N=26) | Delayed Placement (= Control Group) (N=27)
Chest Pains (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient experienced chest pains and went to the hospital emergency room where she was kept overnight to fully evaluate findings. It was determined that she was not having a heart attack but rather gastric reflux
Right knee replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Subject called the day before the surgery to inform us she was having knee replaced the next day.
Bacterial Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Bacterial Pneumonia
Colon Cancer (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject was diagnosed with colon cancer
Hernia surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Surgery to repair hernia
Aortic valve replacement (Cardiac disorders) | 0 (0) | 1 (1) — Patient called on 30-Mar-2018 to inform site he was having aortic valve replacement on 4-APR-2018.
E. Coli (Infections and infestations) | 0 (0) | 1 (1) — Patient reported he was hospitalized with E. coli from June 23-28 with IV antibiotics.
Knee replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — prosthesis knee replacement
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Placement (= Test Group) (N=26) | Delayed Placement (= Control Group) (N=27)
Blisters on my back (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Patient developed painful area on right shoulder. Physician described lesion as ""shingles"" (Herpes Zoster)
Patient stated pain started one week after bridge was placed at #4-#6 on 16NOV2018. Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Bridge removed, surgical intervention on site #5, Bony defect noted at #6d possibly due to resorption at extraction site#5.Debrided and irrigated, sutures placed
Bony defect (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Bridge removed, surgical intervention on site #5, Bony defect noted at #6d possibly due to resorption at extraction site#5.Debrided and irrigated, sutures placed
anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) — After 5 days of amoxicillin, 500mg, patient went to restaurant for seafood. He experienced shortly thereafter lip and faced were swollen and he had difficulty breathing. He went to emergency department (unknown location)
Subject had discomfort around surgical area. (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Intra oral exam shows some irritation around suture on #8 site.
Mass found in ovaries (Reproductive system and breast disorders) | 0 (0) | 1 (1) — patient report mass found in ovaries and it was biopsied. patient did not know results at time of study
Tooth #4 Fractured (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — radiograph taken. Subject give choice of extraction and implant versus RCT and Crown. Subject elected and was scheduled for RCT and Crown
Numbness in face (Nervous system disorders) | 1 (1) | 0 (0) — Patient reported after getting flu shot she got numbness in face, xerostomia, and double vision.
Xerostomia (Nervous system disorders) | 1 (1) | 0 (0) — Patient reported getting Xerostomia after receiving flu shot
Double Vision (Eye disorders) | 1 (1) | 0 (0) — patient had double vision after receiving flu shot
Parathyroid tumor removed (Endocrine disorders) | 1 (1) | 0 (0) — parathyroid tumor removed due to double vision and numbness in face
Nerve Graft Repair (Nervous system disorders) | 1 (1) | 0 (0) — Subject was cutting pineapple and sliced her right thumb. Subject had outpatient nerve repair.
Implant Mobility (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Implant mobile - poor occlusion. Failing dentition with no posterior support.
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Experience vertigo after hernia surgery.
Fracture in right foot and toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Fell and fractured right foot and toe.
Compression Fracture L-1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Compression fracture to L-1 due to a fall
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — Small bowel obstruction resolved on its own.
Salivary stone (mandible) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Subject reports salivary stone, mandibular arch, treated with antibiotics and sour candy.
Right shoulder surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Tendonitis in right shoulder and bicep. Surgery on right shoulder repair tendon.
Small fracture in crown on study tooth (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Small incisal edge porcelain chip on crown of study tooth.
radiolucency around the implant (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Radiolucency around implant at the time of provisional crown delivery. Will follow-up in a week to reevaluate.
implant removed (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Provisional crown was removed and ISQ was 34-35. Implant was mobile and removed. No acute infection was seen (no purulence, edema, or erythema). Granulation tissue was curetted from around the crest of the alveolar ridge and grafted with allograft.
rash on upper chest area possible reaction on antibiotic or mosquito bites (Immune system disorders) | 1 (1) | 0 (0) — on the phone subject complained on redness on the body at the visit: rash visible on upper chest area
infection at implant site with suppuration. Patient came for follow up (Infections and infestations) | 1 (1) | 0 (0) — edema, minimal pus, tenderness on buccal and crestal gingiva but no implant dehiscence inflammation around implant (improved from last visit), edema, erythema buccal and crestal site #9
inflammation around implant (improved from last visit) (Immune system disorders) | 1 (1) | 0 (0) — edema and erythema buccal and crestal site # 9, no purulence
implant came out. Fu S/P removal of failed #9 implant (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — inflammation, edema, erythema, implant is out ST closure achieved. No signs of infection. B-l deficiency present at implant site, will require GBR prior to implant replacement Recommended 4 weeks healing prior to GBR
diagnosis breast cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Not able to complete study procedures due to treatment
Loss of crown (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Loss of cement retention of prosthesis
final screw retained crown delivery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — temporary screw retained crown removed and final screw retained crown delivered
Cold sore (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Subject reported cold sore on upper lip.
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) — Patient had urinary tract infection
Esophageal Tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient was hospitalized for an esophageal tear. He was treated and released.
Worsening high blood pressure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Subject reported an increase in high blood pressure over a period of 9 weeks.
Loose crown (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Subject felt crown loose, but did not fall off. Appointed for the next day, cemented crown removed, and screw retained temporary replaced. New screw retained final crown will be made.
facial implant/fistula (Infections and infestations) | 0 (0) | 1 (1) — patient presented with soft tissue fistula from food impaction. The fistula is not related to the study device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT02569671/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT02569671/SAP_001.pdf